CLINICAL TRIAL: NCT05664022
Title: Effect of Global Postural Reeducation on Low Back Pain Patients With Lower Cross Syndrome. Randomized Controlled Trial
Brief Title: Effect of Global Postural Reeducation on Low Back Pain Patients With Lower Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003923
Record Dates: First submitted 2022-12-12; First posted 2022-12-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain, Postural
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global postural reeducation approach (Experimental): The patient will receive 15 sessions of the Global Postural Re-education approach performed 2times/week for 1 hour including patient education. Each treatment will be individualized for every patient and for his/her pain-related limitation. Each session includes only 2-3 postures to increase the standardization of treatment.
  Interventions: Procedure: Global postural reeducation
- Conventional treatment (Active Comparator): The patient will receive the conventional treatment in form of exercise program of(abdominal and pelvic floor strengthening)and (stretching exercise of back and hip flexor muscles)to improve pain and function in chronic low back pain patients.
  Interventions: Procedure: Global postural reeducation

INTERVENTIONS:
Procedure: Global postural reeducation — The GPR involves a series of active gentle movements and postures aimed at realigning joints, stretching shortened muscles, and enhancing the contraction of antagonist's muscles, thus avoiding postural asymmetry.
  The GPR method includes eight therapeutic postures, lying, sitting or standing, to be held for 15/20 minutes each. Postures can be variously combined during sessions. Postures are chosen on the basis of some parameters, such as the amount of pain, load capacity and age of the patient, and muscle chains to be stretched. to increase the standardization of treatment, it will be proposed only 2 or 3 postures.

SUMMARY:
This study will be conducted toinvestigate the effect of Global Postural Re-education on low back pain patients with Lower cross syndrome

DETAILED DESCRIPTION:
Lower cross syndrome is common, with up to 85% of low back pain cases due to long-term postural faults (Lower crossed syndrome) and it has a negative result on our society. Global Postural Re-education (GPR) is an intervention that is used frequently for chronic low pain to improve pain and function. 50 low back pain patients with lower cross syndrome will be assigned randomly into 2 groups, Group A will receive a Global Postural Re-education approach and consists of 15 treatment sessions of Global Postural Re-education approach, performed 2times/week for 1 hour including patient education. Each treatment is individualized for every patient and for his/her pain-related limitation. Each session includes only 2-3 postures to increase the standardization of treatment. Group B will receive the conventional treatment in form of exercise program of (abdominal and pelvic floor strengthening) and (stretching exercise of back and hip flexor muscles) to improve pain and function in chronic low back pain patients

ELIGIBILITY:
Inclusion Criteria:

* 50 patients.
* Both sexes will be included.
* Patients' age range will be 25 to 40 years old (Esakowitz., 2014).
* Participants will have to meet the criteria for lower crossed syndrome indicating tight hip flexors and erector spinae together with weak glutei and abdominals with low back pain will be presented three months or longer and level of pain intensity more than 3 on VAS.

Exclusion Criteria:

* On other forms of treatment that may interfere with the study including other physical therapy or medication specific to back pain.
* Enrolled in another interventional clinical research trial
* Pregnancy
* Nerve entrapment, bowel or bladder dysfunction and kidney disease.
* Surgery on the back, pelvis or sacrum is indicated or has previously occurred.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
anterior pelvic tilting | up to twelve weeks
  Anterior pelvic tilt will be measured by software application (iHandy Soft, Inc., New York, USA). This application has the capacity to convert the phone into an inclinometer using a built-in sensitive system.It is a tool for assessing angles of slope (or tilt) using all sides of the device plus the camera. A smartphone with the iHandy app can be used in clinical practice and research as an easy and convenient alternative to an inclinometer.
lumbar lordosis | up to twelve weeks
  The lumbar lordosis will be measured by flexible ruler. It is commonly used to measure the degree of spinal curvature of the lumbar lordosis in the sagittal plane. Lumbar lateral X-ray radiography is considered as a golden standard method in lumbar lordosis measurement. However, this method has a number of problems such as being time-consuming and expensive. A flexible ruler is a safe, easy-to-use, and inexpensive tool. Validity between lumbar lordosis measurement with the flexible ruler and the x-ray is 0.91 so the flexible ruler can be used effectively for lumbar lordosis measurements and is a valid, assured, portable and non-invasive tool with high reliability and validity.
flexibility of hip flexors muscle | up to twelve weeks
  Flexibility of hip flexors muscles will be measured by modified Thomas test. This test is performed with the patient supine and the thigh is over the edge of the examining table. The patient is told to grasp the thigh of the untested limb and pull it toward the chest. Lumbar spine is flat on the plinth and the pelvis is in posterior rotation. Length of iliopsoas is determined by measuring the angle of hip ﬂexion. Measurements will be taken pre and post treatment
pain severity | up to twelve weeks
  The pain severity level will be measured via the Visual Analogue Scale (VAS). VAS is a pain rating scale, in which scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10 cm line that represents a continuum between the two ends of the scale "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). In this scale, zero represents the absence of pain, 1-3 shows mild pain, 4-6 denotes moderate pain, and 7-10 indicates severe pain
function disability | up to twelve weeks
  The disability caused by low back pain will be measured via the The Arabic version of Oswestry Low Back Pain Disability Questionnaire. The patient fills out the questionnaire in about 5 minutes and then the doctor scores it in about 1 minute. The patient marks the most relevant answer for each question as accurately as they can. Scoring is done on a scale of 0-5, starting with the first possible answer in the sequence being '0' and the last answer '5'. The maximum possible score for each section is 5. All the scores are added together and divided by the total number of possible points in order to calculate the total score

CONTACTS AND LOCATIONS:
Overall Officials: Enas En Kandil, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour teaching hospital, Damanhūr, Egypt